CLINICAL TRIAL: NCT05495425
Title: Placebo-controlled Comparative Study of NPC-12Y Gel in Patients With Skin Lesions Associated With Tuberous Sclerosis Complex
Brief Title: Clinical Study of NPC-12Y Gel in Patients With Skin Lesions Associated With TSC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPC-12Y-1
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Tuberous sclerosis complex; Sirolimus; Rapalimus gel; mTOR inhibitor
MeSH Terms: conditions — Tuberous Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPC-12Y gel (Experimental): NPC-12Y gel is containing 0.2% Sirolimus
  Interventions: Drug: NPC-12Y gel
- NPC-12Y placebo gel (Placebo Comparator): Placebo gel matched NPC-12Y gel
  Interventions: Drug: NPC-12Y placebo gel

INTERVENTIONS:
Drug: NPC-12Y gel — NPC-12Y gel is applied twice a day for 12 weeks. After the double-blind evaluation period, NPC-12Y gel is applied twice a day for 52 weeks.
  Arms: NPC-12Y gel
Drug: NPC-12Y placebo gel — NPC-12Y placebo gel is applied twice a day for 12 weeks. After the double-blind evaluation period, NPC-12Y gel is applied twice a day for 52 weeks.
  Arms: NPC-12Y placebo gel

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of NPC-12Y gel compared with placebo for skin lesions associated with tuberous sclerosis.

DETAILED DESCRIPTION:
This is a Phase 3, placebo-controlled comparative study of NPC-12Y gel in patients with skin lesions associated with tuberous sclerosis complex. Patients who meet all entry criteria for this study will apply NPC-12Y gel or placebo twice a day for 12 weeks. After the double-blind evaluation period, all patients will apply NPC-12Y gel twice a day for 52 weeks. Approximately 40 eligible patients will be enrolled

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 3 years old or greater at the time of informed consent
2. Patients who are diagnosed as definite diagnosis according to diagnostic criteria for tuberous sclerosis complex (International Tuberous Sclerosis Complex Consensus Conference 2012)
3. Patients with three or more reddish papules of angiofibroma ( >= 2 mm in diameter) on the face at screening tests
4. Patients who are not suitable for therapy with laser or surgery (including liquid nitrogen therapy and phototherapy) for angiofibroma, or who do not want therapy with laser or surgery
5. Patients who are being treated with Rapalimus® gel 0.2% (NPC-12G Gel 0.2%) and who are able to and agree to a withdrawal of at least 4 weeks prior to enrollment in this study.
6. Patients who (or whose guardian) give a written informed consent in understanding and willingness after having received enough explanation regarding the study participation.

Exclusion Criteria:

1. Patients who (or whose guardian) are hard to apply the investigational drug topically with keeping compliance
2. Patients who are hard to be taken pictures of their lesions adequately in such cases that they may not follow instruction of stillness
3. Patients with clinical findings such as erosion, ulcer and eruption on or around the lesion of angiofibroma, which may affect assessment of safety or efficacy
4. Patients with a history or complication of allergy to the component of the investigational drug (sirolimus)
5. Patients who have any infectious disease, cardiac disease, hepatic disease, pulmonary disease, renal disease, hematological disease, or malignant tumor that is considered inappropriate for participation in this clinical study.
6. Patients who have complications such as diseases unsuitable for the trial participation, for examples, uncontrolled diabetes, dyslipidemia, etc.
7. Patients who have participated in other clinical trial or clinical study, and have taken an investigational or clinical study drug within 6 months before the initial registration
8. Patients who used mTOR inhibitors (oral or injectable) other than everolimus within 4 weeks before the initial registration
9. Female patients who are pregnant, may be pregnant, or are lactating
10. Patients who cannot agree to use appropriate contraception after the date of consent to participate in the clinical study and for the duration of the clinical study (including male patients with a partner of childbearing potential)
11. Patients who have received therapy with laser or surgery (including liquid nitrogen therapy and phototherapy) to the lesion of angiofibroma within 6 months before the initial registration
12. Other patients who are considered by the investigator as unsuitable for participation in the clinical study

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Improvements in angiofibroma | 12 weeks
  Improvements comparing with baseline is assessed using photograph by IRC

SECONDARY OUTCOMES:
Improvements in angiofibroma, color and size | 12 weeks
  Improvements comparing with baseline is assessed using photograph by IRC
Index of Facial Angiofibromas (IFA) score | 12 weeks
  Changes in Index of Facial Angiofibromas (IFA) score assessed by investigators

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Gunma University Hospital, Maebashi, Gunma
  - Osaka University Hospital, Suita, Osaka
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - National Hospital Organization Nishi-Niigata Chuo Hospital, Niigata

IPD SHARING:
Plan to Share IPD: No